CLINICAL TRIAL: NCT03911102
Title: A Phase 2a, Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Efficacy, Safety, and Duration of Benefit of Increasing Doses of DaxibotulinumtoxinA for Injection (DAXI for Injection) in the Treatment of Moderate or Severe Lateral Canthal Lines
Brief Title: Efficacy and Safety of Increasing Doses of DaxibotulinumtoxinA for Injection (DAXI for Injection) in the Treatment of Moderate or Severe Lateral Canthal Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1820205
Record Dates: First submitted 2019-03-27; First posted 2019-04-10 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Lateral Canthal Lines
Keywords: Lateral canthal wrinkle; Crow's feet lines; LCL
MeSH Terms: interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: DAXI 12 U (Experimental): DAXI for injection for the treatment of moderate to severe Lateral Canthal Lines (LCL)
  Interventions: Biological: DaxibotulinumtoxinA for injection
- Cohort 2: DAXI 24 U (Experimental): DAXI for injection for the treatment of moderate to severe Lateral Canthal Lines (LCL)
  Interventions: Biological: DaxibotulinumtoxinA for injection
- Cohort 3: DAXI 36 U (Experimental): DAXI for injection for the treatment of moderate to severe Lateral Canthal Lines (LCL)
  Interventions: Biological: DaxibotulinumtoxinA for injection
- Cohort 4: DAXI 48 U (Experimental): DAXI for injection for the treatment of moderate to severe Lateral Canthal Lines (LCL)
  Interventions: Biological: DaxibotulinumtoxinA for injection

INTERVENTIONS:
Biological: DaxibotulinumtoxinA for injection — Intramuscular injection

SUMMARY:
A Phase 2a, Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Treatment of Moderate or Severe Lateral Canthal Lines (LCL).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent consistent with International Conference on Harmonisation (ICH)-Good Clinical Practice (GCP) guidelines and local laws, including authorization to release health information, signed prior to any study procedures being performed
* Be outpatient, male or female subjects, in good general health, 18-65 years old
* Have a score of moderate (2) or severe (3) LCL at maximum smile effort as assessed by the IGA-LCWS
* Able to understand the requirements of the study and be willing and able to follow all study procedures, attend all scheduled visits, and successfully complete the study.

Exclusion Criteria:

* Active skin disease, infections, or inflammation at the injection sites
* History of clinically significant bleeding disorders
* Clinically significant laboratory values at screening that may interfere with a subject's ability to complete the study, as determined by the investigator
* Planned or anticipated need for surgery or hospitalization through the end of the study
* Pregnant, nursing, or planning a pregnancy during the study; or is Women of Child Bearing Potential (WOCBP) but is not willing to use an effective method of contraception
* Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days prior to screening through the end of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Sacramento, CA Site, Sacramento, California
  - Sarasota, FL Site, Sarasota, Florida
  - Itasca, IL Site, Itasca, Illinois
  - Arlington, VA Site, Arlington, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: DAXI 12 U | Cohort 2: DAXI 24 U | Cohort 3: DAXI 36 U | Cohort 4: DAXI 48 U
Started | 15 | 17 | 15 | 16
Completed | 14 | 16 | 12 | 16
Not Completed | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: DAXI 12 U | Cohort 2: DAXI 24 U | Cohort 3: DAXI 36 U | Cohort 4: DAXI 48 U | Total
Number analyzed (Participants) | 15 | 17 | 15 | 16 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 14 | 15 | 61
  >=65 years | 0 | 0 | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 49.9 [34 to 63] | 51.8 [28 to 63] | 52.8 [32 to 65] | 45.5 [27 to 65] | 50 [27 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 13 | 14 | 55
  Male | 1 | 3 | 2 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 0 | 1 | 0 | 1
  Race: Black/African American | 0 | 0 | 0 | 2 | 2
  Race: White | 15 | 16 | 13 | 14 | 58
  Race: Other | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With None or Mild in LCL Severity at Maximum Smile
Description: Percentage of subjects achieving a score or 0 or 1 (none or mild) in LCL severity at maximum smile at Week 4 after LCL treatment on the Investigator Global Assessment Lateral Canthal Wrinkle Severity (IGA-LCWS) scale
Time Frame: Week 4 After LCL Treatment
Population: LCL Evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DAXI 12 U | Cohort 2: DAXI 24 U | Cohort 3: DAXI 36 U | Cohort 4: DAXI 48 U
Number analyzed (Participants) | 15 | 17 | 14 | 16
Participants | 9 | 10 | 8 | 14

ADVERSE EVENTS:
Time Frame: The adverse events were collected throughout the entire study, up to 36 weeks after LCL treatment.
Description: The Safety Population includes all subjects who received at least 1 study treatment injection and was used to assess AEs and SAEs.
Arm/Group | Cohort 1: DAXI 12 U | Cohort 2: DAXI 24 U | Cohort 3: DAXI 36 U | Cohort 4: DAXI 48 U
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/17 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 6/15 | 7/17 | 7/15 | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: DAXI 12 U (N=15) | Cohort 2: DAXI 24 U (N=17) | Cohort 3: DAXI 36 U (N=15) | Cohort 4: DAXI 48 U (N=16)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: DAXI 12 U (N=15) | Cohort 2: DAXI 24 U (N=17) | Cohort 3: DAXI 36 U (N=15) | Cohort 4: DAXI 48 U (N=16)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil percentage increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Center and/or Investigator shall submit to Revance a copy of the proposed publication at least sixty (60) days prior to the submission thereof for publication or disclosure to a third party: (i)to provide Revance with the opportunity to review and comment on the contents thereof, (ii)to identify any Confidential Information to be deleted from the proposed publication or disclosure, and (iii)or delay the publication or disclosure 90 days to allow Revance to pursue patent protections.

DOCUMENTS (2):
  • Study Protocol (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT03911102/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03911102/SAP_001.pdf